CLINICAL TRIAL: NCT05385328
Title: Multisensorial Analysis of Human Activity for Diagnosis and Early Detection of Functional Limitations (EYEFUL)
Brief Title: Multisensorial Analysis of Human Activity for Diagnosis and Early Detection of Functional Limitations
Acronym: EYEFUL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nuria Máximo-Bocanegra (Other)
Collaborators: AlcaládeHenaresU (Unknown)
Responsible Party: Sponsor-Investigator, Nuria Máximo-Bocanegra, Occupational Therapist Philosophy Doctor (PhD) (team investigator), Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Other Study IDs: KingJuanCarlosU
Record Dates: First submitted 2022-02-21; First posted 2022-05-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2022-11

CONDITIONS: Handicaps Physical; Fetal Alcohol Syndrome; Mental Disability
Keywords: Activities of Daily Life; Clinical evaluation; Multisensorial analysis
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy people: Undiagnosed persons will be evaluated by the EYEFUL system performing activities of daily living. Patterns of action will be recorded, to establish outcome measures in healthy population.
  Interventions: Device: EYEFUL: healthy people
- people with physical or psychological diagnoses: People with various clinical diagnoses will be evaluated by the EYEFUL system performing activities of daily living. Patterns of action will be recorded, in order to establish outcome measures in comparison with healthy population and with other diagnoses.
  Interventions: Device: EYEFUL: people with pathology

INTERVENTIONS:
Device: EYEFUL: healthy people — This kind of study implies that we do not require the use of any substance, medicine or therapeutic technique and neither imply any risk to the participants.
  The data to be captured are exclusively video and audio recordings, and different signals from smart watches (mainly related to movement). Addittionaly, the clinical evaluation of the performance of these activities will be carried out according to the assessment scales to be defined in the project. The results of this evaluation will be exclusively used in the training of the automatic systems developed in the project and in order to establish a correlation between the captured observations (video, audio, smart watches signals) and the diagnostic assessment.
  Groups: Healthy people
Device: EYEFUL: people with pathology — This kind of study implies that we do not require the use of any substance, medicine or therapeutic technique and neither imply any risk to the participants.
  The data to be captured are exclusively video and audio recordings, and different signals from smart watches (mainly related to movement). Addittionaly, the clinical evaluation of the performance of these activities will be carried out according to the assessment scales to be defined in the project. The results of this evaluation will be exclusively used in the training of the automatic systems developed in the project and in order to establish a correlation between the captured observations (video, audio, smart watches signals) and the diagnostic assessment.
  Groups: people with physical or psychological diagnoses

SUMMARY:
Physical and cognitive changes provoked by a pathology worsen the functional capability of the individual making it more difficult to perform Activities of Daily Living (ADLs) and causing dependency and/or disability. There are standardized observational tests for the clinical assessment of the degree of functional limitation in basic or instrumental ADLs (e.g., Assessment Motor and Process Skills - AMPS). On the other hand, all these tests bear the problem of the subjectivity of the evaluator in the analysis. The presence of the evaluator in the test may have an influence in the way a subject performs ADLs.

The goal of the project is to develop a methodology to design, implement and validate automatic clinical tests of functional limitation, that: 1) give objective assessments with clinical validity, and 2) remove the interference in the test execution caused by the physical presence of the evaluator.

DETAILED DESCRIPTION:
Physical and cognitive changes provoked by a pathology worsen the functional capability of the individual making it more difficult to perform Activities of Daily Living (ADLs) and causing dependency and/or disability. There are standardized observational tests for the clinical assessment of the degree of functional limitation in basic or instrumental ADLs (e.g., Assessment Motor and Process Skills - AMPS). On the other hand, all these tests bear the problem of the subjectivity of the evaluator in the analysis. The presence of the evaluator in the test may have an influence in the way a subject performs ADLs.

The goal of the project is to develop a methodology to design, implement and validate automatic clinical tests of functional limitation, that: 1) give objective assessments with clinical validity, and 2) remove the interference in the test execution caused by the physical presence of the evaluator. The human evaluator subjectivity will be replaced with an automatic system that extracts multimodal (i.e., multisensorial) information from the environment during the user functional assessment. Specifically including audio, video and depth sensors and the information collected from wearable sensors that the subject under test may carry. The objective assessment will also provide clues that, given the subject clinical history, can be used for early detection of limitations.

This problem has not been systematically addressed in the literature. The project is thus a first solution of the development and clinical validation of an automated system that allows an objective evaluation of observational tests. Tackling the clinical assessment of functional limitations will be then performed in an adapted real environment (equipped with the adequate electronic sensors) in the URJC facilities.

The EYEFUL-URJC subproject has a key role in the methodological design and clinical validation of the automatic evaluation tools. They will also carry out the actual tests over normal subjects and patients comparing the output of the current tools, as AMPS, with the output of the assessment tools developed for the project. In order to extract relevant features from video, depth, audio and other sensors, the project leverages the research experience on automatic sensing of human activities in intelligent spaces of EYEFUL-UPM and EYEFUL-UAH. The EYEFUL-UPM subproject concentrates in the analysis of the subject face, head pose, gaze, and accurate 3D alignment of the facial landmarks, that enable the estimation facial attributes useful for different tests (i.e., focus of attention, presence of pain, confusion, fear, etc.). The EYEFUL-UAH subproject concentrates the analysis on the user whole body activity and her/his interaction with objects, with depth and video sensors, and integrating also audio and wearables' data to automatically assess the functional capability of the evaluated persons. The three coordinated groups approach the project in an interdisciplinary way, with strong feedback requirements among them all along the development. This close interaction is fundamental to ensure the adequate focus of the technical developments given the strict clinical requirements of the task.

ELIGIBILITY:
Inclusion criteria:

* People with a Certificate of Disability from the Ministry of Health, Consumer Affairs and Welfare.
* Degree of disability (percentage from 0-90%, where 100% reflects the maximum disability)
* over 18 years of age.

Exclusion criteria:

* Inability to follow-2-step commands.
* If participant is unwilling to travel for assessment.
* Currently in treatment with: Psychotropics, Antipsychotics and/or Benzodiazepines.
* People with a Certificate of Disability from the Ministry of Health, Consumer Affairs and Welfare.
* Degree of disability (percentage of 90-100%, where 100% reflects the maximum disability)
* Refusal to sign the informed consent form.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control group sample will be obtained by convenience, through the contacts of the research group and the university environment. In turn, a group of subjects with a medical diagnosis will be selected from the Hospital Universitario Fundación Alcorcón and the Hospital Universitario Ramón y Cajal of the Community of Madrid.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Physical measures | Frist year
  These measures of the subject's physical condition shall be monitored while the subject is performing the assessment activities. This measure is heart rate measured in beats per minute.
Physical measures 2 | Frist year
  These measures of the subject's physical condition shall be monitored while the subject is performing the assessment activities. This measure is oxygen saturation expressed as a percentage.
Accelerometry | Frist year
  Accelerometers will be used to measure energy expenditure expressed in METs.
Accelerometry 2 | Frist year
  Accelerometers will be used to measure walking speed in metres per second.
Accelerometry 3 | Frist year
  Accelerometers will be used to measure displacement or distance travelled in metres.
Facial expression | second year
  Collected through the Observed Emotion Rating Scale (OERS), this is an observational measure with 6 types of emotions, 3 positive (pleasure, interest, satisfaction) and three negative (sadness, anxiety and anger). This scale is to be performed after a 10-minute observation. The scores are the observers' estimates of the amounts of time, during the 10-minute interval, that each emotion was exhibited: Never, < 16 sec, 15-59 sec, 1-5 min, > 5 min, and "can't say".
Quality of performance | second year
  This is assessed using the standardised tool "Assessment of Motor Process Skills (AMPS)". It measures the quality of performance of tasks related to activities of daily living (ADL) in a natural environment. It is a tool designed to measure the interaction between the person, the ADL task and the environment.
Functional ability | second year
  An assessment questionnaire known as the "Activities of Daily Living Questionnaire (ADLQ)" will be used. It measures a subject's functional ability and performance in 6 areas, which allow for a complete profile of deficits related to daily functioning. The final scores are calculated with a specific formula that provides a percentage of functional impairment from 0 to 100. There are total scores and scores per subscale.
Severity of anxiety and depression | second year
  The Hamilton Anxiety Rating Score (HARS) is used to measure the severity of anxiety in a global way in subjects with anxiety or depression. In addition, this instrument is useful for monitoring response to treatment. It is a heteroadministered tool and the total score is the sum of each of the items, the range of scores being between 0 and 56.
Self-perception of performance | second year
  The Canadian Occupational Performance Measure (COPM) is a semi-structured interview that allows for a dialogue between the patient and the assessor, designed to measure the patient's self-perception of performance in daily life. It assesses 3 areas: Self-care, Productivity (or work) and Leisure. Within each area, psychological, physical, socio-cultural and spiritual components are analysed, in addition to the performance and satisfaction linked to the performance of the activities. The total score will be an arithmetic mean for the performance value and another for satisfaction, the range can be from 1 to 10 and higher scores indicate better levels of performance and high satisfaction with performance.
Functional cognitive performance | second year
  The Kettle Test is a performance test designed to indicate a person's ability to perform everyday tasks. The clinician observes while the subject completes the task, which involves making two hot drinks, one for the assessor and one for the subject. Performance is assessed and scores are based on 13 performance indices. Items are scored from 0 to 4. The score can be as high as 52, with higher scores revealing more severe performance problems.
Cognitive processing | second year
  The Allen Cognitive Level Screen-5 (ACLS-5) is a measurement instrument established in the theoretical context of the cognitive impairment model, created by Claudia Allen.
  It is used to obtain rapid information about global cognitive processing capacity, learning potential and performance abilities and to detect unknown or suspected problems related to functional cognition.
Degree of disability and quality of life | second year
  To measure the degree of disability, the WHO Disability Assessment Scale, WHO-DAS 2.0 (WD2), measures changes in functioning and their levels of difficulty in performing and carrying out daily activities. The WD2 scale is composed of 36 items divided into 6 domains, assessed through a Likert scale with values from 1 to 5, referring to the difficulty presented. Higher scores indicate a greater degree of disability. The total score ranges from 36-180.
Analytical validation | Third year
  This step moves the evaluation procedure of EYEFUL sensors from the sensor itself (algorithm) to in vivo (evaluates on the person). In this phase, the data converts the sensor measurements into physiological metrics. The sensor measurements are compared with the Gold Standard scales mentioned above. Subsequently, an analysis of the convergent validity of the assessments will be made. Finally Eyeful, could be used to assess functional capabilities in a sample of subjects recruited with pathology to demonstrate that the developed systems acceptably identify, measure or predict functional status or experience in the defined context

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad Ciencias de la Salud. Universidad Rey Juan Carlos, Madrid, Alcorcón, Spain

IPD SHARING:
Plan to Share IPD: No
No personal data of participants will be shared